CLINICAL TRIAL: NCT03392974
Title: A Phase 3 Open-Label, Single-Arm Study To Evaluate The Efficacy and Safety of BMN 270, an Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII at a Dose of 4E13vg/kg in Hemophilia A Patients With Residual FVIII Levels ≤1IU/dL Receiving Prophylactic FVIII Infusions
Brief Title: Single-Arm Study To Evaluate The Efficacy and Safety of Valoctocogene Roxaparvovec in Hemophilia A Patients at a Dose of 4E13 vg/kg
Acronym: GENEr8-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 270-302; 2017-003573-34 (EudraCT Number)
Record Dates: First submitted 2017-12-22; First posted 2018-01-08 (Actual); Results first posted 2021-10-08 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; Gene Therapy; Clotting Disorders; Blood Disorder; Blood Coagulation Disorders; Inherited Blood Coagulation Disorders; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases; Inborn; Factor VIII; Coagulants
MeSH Terms: conditions — Hemophilia A; Hemostatic Disorders; Hematologic Diseases; Blood Coagulation Disorders; Blood Coagulation Disorders, Inherited; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn | interventions — Valoctocogene Roxaparvovec

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Valoctocogene Roxaparvovec Open Label (Experimental): Single administration of valoctocogene roxaparvovec at a dose of 4E13 vg/kg
  Interventions: Biological: Valoctocogene Roxaparvovec

INTERVENTIONS:
Biological: Valoctocogene Roxaparvovec — Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Hemophilia A
  Other Names: BMN 270

SUMMARY:
This Phase III clinical study will assess the efficacy of BMN 270 defined as FVIII activity, during weeks 49-52 following intravenous infusion of BMN 270 and assess the impact of BMN 270 on usage of exogenous FVIII replacement therapy and the number of bleeding episodes from week 5 to week 52.

ELIGIBILITY:
Inclusion Criteria:

1. Males ≥ 18 years of age with hemophilia A and residual FVIII levels ≤ 1 IU/dL as evidenced by medical history.
2. Must have been on prophylactic FVIII replacement therapy for at least 12 months prior to study entry.
3. Treated/exposed to FVIII concentrates or cryoprecipitate for a minimum of 150 exposure days.
4. No previous documented history of a detectable FVIII inhibitor of less than 0.6 Bethesda Units (BU).

Exclusion Criteria:

1. Detectable pre-existing antibodies to the AAV5 capsid.
2. Any evidence of active infection or any immunosuppressive disorder, including HIV infection.
3. Significant liver dysfunction, prior liver biopsy showing significant fibrosis, liver cirrhosis of any etiology or history of hepatic malignancy.
4. Evidence of any bleeding disorder not related to hemophilia A.
5. Active Hepatitis C.
6. Prior treatment with any vector/gene transfer agent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological males only
Enrollment: 1 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2023-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (1):
- Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- BMN 270 4E13 vg/kg: Single administration of valoctocogene roxaparvovec at a dose of 4E13 vg/kg
Period: Overall Study
Arm/Group | BMN 270 4E13 vg/kg
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BMN 270 4E13 vg/kg
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (NA) — The number of participants is 1, so the Standard Deviation is Not Applicable.
Age, Customized [Number; unit: participants]
  18 - <65 | 1
  >= 65 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  Other | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Change of the Median Factor VIII (FVIII) Activity
Description: Change of the FVIII activity, as measured by chromogenic substrate assay, at Week 52 post-BMN 270 infusion.
Time Frame: Week 52
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | BMN 270 4E13 vg/kg
Number analyzed (Participants) | 1
IU/dL | 4.1 (NA) — The number of participants is 1, so the Standard Deviation was not calculated

2. Secondary Outcome: Change in the Annualized Utilization (IU/kg) of Exogenous FVIII Replacement Therapy
Description: Change in the annualized utilization (IU/kg) of exogenous FVIII replacement therapy during Week 5 to Week 52 post-BMN 270 infusion from the baseline utilization of exogenous FVIII replacement therapy
Time Frame: Weeks 5 through Week 52
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: IU/kg/yr
Arm/Group | BMN 270 4E13 vg/kg
Number analyzed (Participants) | 1
IU/kg/yr | -4058.24 (NA) — The number of participants is 1, so the Standard Deviation was not calculated

3. Secondary Outcome: Change in the Annualized Number of Bleeding Episodes Requiring Exogenous FVIII Replacement Treatment
Description: Change in the annualized number of bleeding episodes requiring exogenous FVIII replacement treatment (annualized bleeding rate, ABR) during Week 5 to Week 52 of the study post-BMN 270 infusion from the baseline ABR
Time Frame: Weeks 5 though Week 52
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: episodes/year
Arm/Group | BMN 270 4E13 vg/kg
Number analyzed (Participants) | 1
episodes/year | 5.77 (NA) — The number of participants is 1, so the Standard Deviation was not calculated

ADVERSE EVENTS:
Time Frame: First 52 weeks post infusion
Groups:
- Total: Total
Arm/Group | BMN 270 4E13 vg/kg | Total
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 270 4E13 vg/kg (N=1) | Total (N=1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 1 (2) | 1 (2)
Nasopharyngitis (Infections and infestations) | 1 (4) | 1 (4)
Alanine aminotransferase increased (Investigations) | 1 (4) | 1 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT03392974/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT03392974/SAP_001.pdf